CLINICAL TRIAL: NCT06027632
Title: Remotely Supervised Computerized Cognitive Stimulation to Reduce Post-chemotherapy Cognitive Difficulties in Patients Treated for Localized Breast Cancer: a Multicenter Randomized Controlled Trial
Brief Title: Remotely Supervised Computerized Cognitive Stimulation to Reduce Post-chemotherapy Cognitive Difficulties in Patients Treated for Localized Breast Cancer
Acronym: COG STIM 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-A01134-41
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Cognitive Dysfunction
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction | interventions — Organization and Administration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remotely-supervised online cognitive stimulation intervention (Other)
  Interventions: Other: Cognitive exercises with supervision
- Open access to online home-based cognitive exercises without supervision (Other)
  Interventions: Other: Cognitive exercises without supervision

INTERVENTIONS:
Other: Cognitive exercises with supervision — The experimental group will receive a 12-week intervention consisting of three 20-minute online cognitive stimulation sessions per week along with a weekly 30-minute centralized online remote supervision session with a neuropsychologist. Patient will also have access to the "PRESCO" program of the "HAPPYNeuron-Pro" software, which is designed to train up to 12 different cognitive domains, including attention, memory, executive functions and processing speed
  Arms: Remotely-supervised online cognitive stimulation intervention
Other: Cognitive exercises without supervision — Patient will have access to the program named "PRESCO" of the "HAPPYNeuron-Pro" software, which is designed to train up to 12 different cognitive domains, including attention, memory, executive functions and processing speed
  Arms: Open access to online home-based cognitive exercises without supervision

SUMMARY:
Investigator propose the first French randomized comparative study to assess the efficacy of a remotely supervised online cognitive stimulation program, compared to an unsupervised online cognitive exercise intervention, in reducing cognitive complaints in localized breast cancer patients after adjuvant chemotherapy. Previous randomized studies have confirmed the effectiveness of online cognitive stimulation programs compared to standard care. The study seeks to determine the added value of remote supervision by a neuropsychologist. The control group will have access to the same online cognitive exercises as the experimental group but without supervision. Investigator has chosen not to include a wait-list group as it would be unethical to deny patients with cognitive complaints the opportunity to participate in an intervention expected to benefit them. The secondary objective is to evaluate the benefit of the supervised digitalized cognitive intervention on objective cognitive impairment.

The research hypothesis is that incorporating personalized remote support with supervision from a neuropsychologist into a digitalized cognitive stimulation program will reinforce the effectiveness of the intervention on cognitive complaints. This will be achieved by improving participation/adherence to the online cognitive stimulation program, as well as through the personalized supervision itself. Investigator believe that the supervision sessions, including educational components, will enable patients to identify their strengths, promote their cognitive awareness, and develop individualized strategies to apply their compensatory abilities in real-life situations. Since cognitive difficulties have multiple underlying causes, reducing these symptoms requires a multifaceted approach. The hypothesis is that combining cognitive training (which increases neuroplasticity and directly targets the cognitive domains affected by cancer and its treatments), with structured supervised educational sessions based on compensatory strategies, will yield better outcomes than online cognitive stimulation alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with localized breast cancer
* Age 18 or older,
* Who have received adjuvant or neo-adjuvant chemotherapy and are currently undergoing adjuvant radiotherapy (ongoing hormone therapy, maintenance therapy other as target therapies or immunotherapy are permitted) until 6 months after end of radiotherapy.
* Patients who report cognitive complaints that significantly impact their quality of life, as evaluated by the quality of life subscale of the FACT-Cog questionnaire. This subscale is composed by 4 questions:

  1. I have been upset about these problems;
  2. These problems have interfered with my ability to work;
  3. These problems have interfered with my ability to do things I enjoy;
  4. These problems have interfered with the quality of my life.

Patients are eligible if their score on this subscale is at or below the 10th percentile, based on age guidelines and normative data (Lange et al., 2015), namely:

* ≤ 8 for patients aged 30-49 years
* ≤ 9 for patients aged 50-69 years
* ≤ 10 for patients aged 70-89 years

  * Patients who have completed at least three years of primary school education, as determined by the Barbizet scale,
  * Patient with access to a functional laptop/computer with a keyboard, internet connection and an e-mail account - being able to use those tools alone,
  * Fluent in French,
  * Patients who have provided informed consent to participate in the study.

Exclusion Criteria:

* Personality disorder or any known progressive psychiatric pathology (e.g. schizophrenia),
* Previous neurological history with ongoing cognitive symptoms (sequelae of head trauma, stroke, multiple sclerosis, epilepsy, neurodegenerative pathology, etc.),
* Excessive alcohol intake or drug use, which could compromise participation to the intervention
* Major visual and/or hearing deficit,
* Patient who might not be able to complete neuropsychological testing, (including those with significant cognitive disorders that impede the completion of cognition tests, as determined by the cognitive screening test MoCA (MONTREAL COGNITIVE ASSESSMENT) and based on age and educational level according to GRECOGVASC (Reflection Group for Vascular COGnitive Assessment) normative data)
* Already participating in a cognitive training program,
* Refusal to participate,
* Patient deprived of liberty or under guardianship,
* Patient who might not be able to participate due to geographic, social or psychopathological reasons.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Average change in the score of the Perceived Cognitive Impairment (PCI) subscale score of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | After 12 weeks
  Perceived Cognitive Impairment (PCI) score range 0-72 (The higher the score, the fewer cognitive complaints)

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre hospitalier de Bligny, Briis-sous-Forges
  - Centre François Baclesse, Caen
  - CH Métropole Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Hôpital privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Clinique Haute Energie, Nice
  - CHU de Nimes, Nîmes
  - Hôpital Saint-Louis, Paris
  - La Pitié Salpétrière, Paris
  - Centre hospitalier de Pau, Pau
  - Centre Arrmoricain d'Oncologie, Plérin
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - Clinique Medico-chirurgicale Charcot, Sainte-Foy-lès-Lyon
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bousquet M, Lange M, Lequesne J, Durand-Zaleski I, Diaz O, Di Meglio A, Bachelot T, Grellard JM, Clarisse B, Joly F. Remotely supervised online cognitive training to reduce cognitive difficulties following chemotherapy in patients treated for localized breast cancer: Protocol of the Cog-Stim2 multicenter randomized controlled trial. PLoS One. 2025 Nov 13;20(11):e0335124. doi: 10.1371/journal.pone.0335124. eCollection 2025. PMID 41231878